CLINICAL TRIAL: NCT06086223
Title: Functional Outcomes Following Ankle Fracture Fixation With or Without Ankle Arthroscopy: Randomized Control Study
Brief Title: Functional Outcomes Following Ankle Fracture Fixation With or Without Ankle Arthroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, El-Taher Alaa Eldin Ahmed Eid, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Arthroscopy for ankle fracture
Record Dates: First submitted 2023-10-07; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Ankle Fractures; Ankle Injuries; Arthroscopic Surgery
Keywords: functional outcomes of ankle fracture management; ankle scope; syndesmosis reduction; ankle ligaments evaluation
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries | interventions — Arthroscopy

STUDY DESIGN:
Intervention Model Description: Based on determining outcome variable, the estimated minimum required sample size is 176 cases (88 cases in each group).
  The sample size was calculated using G*power software 3.1.9.7., based on the following assumptions: the patient satisfaction rate was higher in those patients who underwent arthroscopy compared with ORIF alone (93% vs 75%, P ¼ .05) (5).
  Main statistical test is z test, Alpha = 0.05, Power = 0.95 Allocation ratio= 1.
Who Masked: Outcomes Assessor
Masking Description: Random assignment of intervention will be done after subjects have been assessed for eligibility and recruited. The sealed opaque envelope method will be used for randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- those patients who will go for ORIF plus arthroscopy (Experimental): we will start with a standard ankle arthroscopy. A leg holder and ankle joint distractor will be used. We will start with the anteromedial portal and introduce the 4-mm scope into the ankle joint. Next, under direct visualization, and taking care to preserve any branches of the superficial peroneal nerve, we will perform the anterolateral portal.
  We will carry out a standard diagnostic ankle arthroscopy to evaluate the ankle cartilage, wash intra-articular haematoma, identify, and remove any intra-articular fracture fragments and loose bodies, perform dynamic ligamentous stress examinations while directly visualizing the syndesmosis, the deltoid ligament, and the lateral collateral ligament.
  Following fracture fixation, arthroscopy will be also used as a second look to evaluate the quality of both articular and syndesmotic reduction, perform any needed arthroscopic intervention for deltoid ligament injury or management of chondral lesions (OCLs)
  Interventions: Procedure: ankle arthroscopy with ORIF
- patients who will go for ORIF without arthroscopy (Experimental): * Posterior malleolus fractures will be addressed when it is present whatever its size.
  * The fibula fractures will be fixated using either a posterolateral or direct lateral incision. Lag screws will be used when the fracture pattern allows, and all fractures will be also treated with a neutralization or antiglide plate depending on the pattern and approach.
  * If a medial malleolus fracture is present, this will be addressed through a direct medial incision. These fractures will be either fixed with cannulated screws or tension band cerclage wiring or a plate and screw construct depending on the fracture pattern.
  * Once all bony injuries will be stabilized, a Cotton test will be performed under live fluoroscopy to determine syndesmosis stability. If positive, the syndesmosis will be stabilized using fully threaded screws.
  Interventions: Procedure: fracture ankle fixation without ankle arthroscopy

INTERVENTIONS:
Procedure: ankle arthroscopy with ORIF — we will go for fixation of the fracture with association of scope intervention pre and post fixation
  Other Names: ankle fracture fixation with arthroscopy
  Arms: those patients who will go for ORIF plus arthroscopy
Procedure: fracture ankle fixation without ankle arthroscopy — we will go for fixation of the fracture alone with no scope intervention
  Other Names: ankle fracture fixation without arthroscopy
  Arms: patients who will go for ORIF without arthroscopy

SUMMARY:
The aim of our study is to identify if there is statistically significant difference in patient reported functional outcomes in cases of unstable ankle fracture managed by ORIF with and without ankle arthroscopy.

DETAILED DESCRIPTION:
Acute ankle fracture is one of the commonest fractures of the lower limb. Anatomical reduction and stable fixation remain the main surgical treatment for unstable ankle fractures . However, its final outcomes are not as good as expected . Fracture malunion, failure to address the disrupted syndesmosis and associated ligamentous or chondral lesions can be reasons for poor surgical outcome.

1-mm of lateral talar shift lead to a 42% increase in contact stress, so the anatomic reduction is critical to the long-term integrity of the joint . It is difficult to assess 1 to 2 mm of mal-reduction with C-arm fluoroscopy. The best assessment of the syndesmotic reduction is performed with axial CT imaging of the ankle.

Ankle arthroscopy is expected to be a more sensitive tool for syndesmotic disruption diagnosis and other intra-articular pathologies and as a guide for anatomical reduction of the syndesmosis . Several studies have reported the incidence of chondral lesions seen during ankle arthroscopy at the time of ankle fracture ORIF, but those studies report the role of arthroscopy as a diagnostic or predictive tool for patient outcome. Very few studies have discussed the rates of arthroscopic intervention, the procedures performed, and the association of these procedures with patient final functional outcomes .

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥16 years of age who will be managed operatively for:

  * rotational ankle fracture Danis-Weber classification B or C fibula fracture
  * fracture dislocation ankle
  * Fractures extending into the tibial plafond,
  * Talus fractures (body or neck) in our institution

Exclusion Criteria:

Pediatric fractures, Polytrauma patients, Fractures managed with closed-contact casting and, patients with lost follow up during this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Society(AOFAS) hindfoot score | 6 months and one year follow up
  AOFAS hindfoot score difference between the 2 groups at 6 months and one year postoperatively from 0 to 100 where higher value indicates better functional outcomes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith KS, Drexelius K, Challa S, Moon DK, Metzl JA, Hunt KJ. Outcomes Following Ankle Fracture Fixation With or Without Ankle Arthroscopy. Foot Ankle Orthop. 2020 Mar 2;5(1):2473011420904046. doi: 10.1177/2473011420904046. eCollection 2020 Jan. PMID 35097364
- [Background] Zengerink M, Struijs PA, Tol JL, van Dijk CN. Treatment of osteochondral lesions of the talus: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2010 Feb;18(2):238-46. doi: 10.1007/s00167-009-0942-6. Epub 2009 Oct 27. PMID 19859695